CLINICAL TRIAL: NCT03963011
Title: Pilot Randomized Control Trial of Necrotizing Enterocolitis Screening Abdominal Radiograph Versus Bowel Ultrasound Plus Abdominal Radiograph in Premature Neonates
Brief Title: NEC Screening Abdominal Radiograph vs Bowel Ultrasound in Preemies
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low Recruitment
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 17030157
Record Dates: First submitted 2018-12-19; First posted 2019-05-24 (Actual); Results first posted 2022-01-10 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2021-12

CONDITIONS: Enterocolitis, Necrotizing; Premature Infant
Keywords: NEC; Necrotizing Enterocolitis; Premature Infant; Calprotectin
MeSH Terms: conditions — Enterocolitis, Necrotizing; Premature Birth

STUDY DESIGN:
Intervention Model Description: Infants randomized to the AXR only arm will obtain an AXR as per standard of care. Repeat AXR, if any, will be left to the discretion of the treating neonatologist. In this arm, no BUS study will be performed unless the attending neonatologist decides it is clinically indicated. This situation is expected to be exceedingly rare, as BUS is not part of the standard of care for NEC evaluation. Infants randomized to the AXR and BUS arm will also get an AXR, with repeat AXR left to the discretion of the treating neonatologist. In addition to this standard of care, infants randomized to this arm will receive a BUS as the intervention. This BUS will be ordered at the same time as the initial AXR and will be performed within six hours of the order being placed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Arm A: AXR Only (No Intervention): Infants randomized to Arm A will obtain an abdominal x-ray (AXR) as per standard of care
- Arm B: AXR + Bowel US (Active Comparator): Infants randomized to Arm B will obtain an abdominal x-ray (AXR) as per standard of care and a bowel ultrasound (BUS) as the intervention
  Interventions: Diagnostic Test: Bowel Ultrasound

INTERVENTIONS:
Diagnostic Test: Bowel Ultrasound — Ultrasound imaging of the bowel
  Arms: Arm B: AXR + Bowel US

SUMMARY:
The overall primary objective is to establish the feasibility and pilot the design and delivery of a diagnostic randomized controlled trial (RCT) of BUS (bowel ultrasound) for NEC evaluation which will lead to a successful application for a larger, multi-center clinical trial in the future. This program of research is anticipated to have a significant positive impact in the timely and accurate diagnosis of NEC in preterm infants.

DETAILED DESCRIPTION:
Necrotizing enterocolitis (NEC) is the most common bowel disease in premature and low birth weight neonates. NEC is defined by the loss of mucosal integrity of the bowel wall enabling bacteria and other toxins to permeate into the bowel causing ischemia and necrosis which can lead to bowel perforation and sepsis. NEC can result in substantial morbidity and mortality and prolonged hospital stay.

In the past, abdominal radiography has been scored on a standard scale that correlated with outcomes. Duke University Medical Center developed a standardized ten-point radiographic scale, the Duke Abdominal Assessment Scale (DAAS) (Appendix B) and was proven to be directly proportional to the severity of NEC on patients that underwent surgery. Abdominal radiographs are assessed for gas pattern, bowel distention, location and features, pneumatosis (gas in bowel wall), portal venous gas, and pneumoperitoneum (free air in peritoneal cavity) to indicate the level of suspicion of NEC. The use of abdominal radiographs is the most common assessment for suspected NEC in infants, however, there have been recent studies done on the utility of bowel ultrasound to aid in early diagnosis of NEC due to the ability to evaluate peristalsis, echogenicity and thickness of bowel wall, pneumatosis and the capability of doing color Doppler to evaluate blood perfusion. A University of Toronto study used ultrasound to assess bowel perfusion with color Doppler in neonates and found a correlation between absence of bowel wall perfusion and the increased severity of NEC on surgical pathology. Although there are similar signs found between abdominal radiography and bowel ultrasound, some of the more severe features such as, pneumoperitoneum, were found to be more sensitive on bowel ultrasound, thus potentially leading to more definitive treatment. Currently, there is no good study evaluating whether the use of bowel ultrasound affects clinical outcomes in VLBW patients over the use of abdominal radiography alone.

The use bowel ultrasound has yet to be adopted in the setting of suspicion for NEC at our institution. This is primarily due to the lack of expertise of the ultrasound technologists, radiologists and clinicians. With literature dating back to 2005 supporting the use of bowel ultrasound in diagnosis of severity of NEC, we would like to see if a regimen involving combined ultrasound and radiograph screening for NEC would make a difference in clinical outcomes (morbidity, mortality, and length of stay (LOS)) compared with radiograph screening alone.

Calprotectin is a protein found in the stool that, at elevated levels, indicates gastrointestinal inflammation. The addition of fecal biomarkers to the diagnostic work up for NEC also has promising impact. It has been suggested that fecal calprotectin levels obtained at the time of suspicion of NEC may be a useful noninvasive indicator to determine the severity of inflammation in the intestine and whether it is related to NEC or other forms of inflammation. Correlation of the fecal biomarkers with findings on BUS may be helpful to more definitively diagnose NEC.

ELIGIBILITY:
Inclusion Criteria:

* • Neonates born prior to or at 28 weeks gestation admitted to NICU at CMH

Exclusion Criteria:

* Infants with chromosomal or multiple congenital anomalies
* Unable to ultrasound the bowel (e.g. gut in silo, omphalocele, gastroschisis)
* Infants who are greater than 36 corrected weeks upon admission

Max Age: 28 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Actual)
Dates: Start 2018-12-20 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erin Opfer, DO, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Epelman M, Daneman A, Navarro OM, Morag I, Moore AM, Kim JH, Faingold R, Taylor G, Gerstle JT. Necrotizing enterocolitis: review of state-of-the-art imaging findings with pathologic correlation. Radiographics. 2007 Mar-Apr;27(2):285-305. doi: 10.1148/rg.272055098. PMID 17374854
- [Background] Staryszak J, Stopa J, Kucharska-Miasik I, Osuchowska M, Guz W, Blaz W. Usefulness of ultrasound examinations in the diagnostics of necrotizing enterocolitis. Pol J Radiol. 2015 Jan 1;80:1-9. doi: 10.12659/PJR.890539. eCollection 2015. PMID 25574248
- [Background] Coursey CA, Hollingsworth CL, Gaca AM, Maxfield C, Delong D, Bisset G 3rd. Radiologists' agreement when using a 10-point scale to report abdominal radiographic findings of necrotizing enterocolitis in neonates and infants. AJR Am J Roentgenol. 2008 Jul;191(1):190-7. doi: 10.2214/ajr.07.3558. PMID 18562745
- [Background] Coursey CA, Hollingsworth CL, Wriston C, Beam C, Rice H, Bisset G 3rd. Radiographic predictors of disease severity in neonates and infants with necrotizing enterocolitis. AJR Am J Roentgenol. 2009 Nov;193(5):1408-13. doi: 10.2214/AJR.08.2306. PMID 19843760
- [Background] Faingold R, Daneman A, Tomlinson G, Babyn PS, Manson DE, Mohanta A, Moore AM, Hellmann J, Smith C, Gerstle T, Kim JH. Necrotizing enterocolitis: assessment of bowel viability with color doppler US. Radiology. 2005 May;235(2):587-94. doi: 10.1148/radiol.2352031718. PMID 15858098
- [Background] Kim WY, Kim WS, Kim IO, Kwon TH, Chang W, Lee EK. Sonographic evaluation of neonates with early-stage necrotizing enterocolitis. Pediatr Radiol. 2005 Nov;35(11):1056-61. doi: 10.1007/s00247-005-1533-4. Epub 2005 Aug 3. PMID 16078076
- [Background] Nakayuenyongsuk W, Christofferson M, Stevenson DK, Sylvester K, Lee HC, Park KT. Point-of-Care Fecal Calprotectin Monitoring in Preterm Infants at Risk for Necrotizing Enterocolitis. J Pediatr. 2018 May;196:98-103.e1. doi: 10.1016/j.jpeds.2017.12.069. Epub 2018 Mar 6. PMID 29519542
- [Derived] Cuna A, Chan S, Jones J, Sien M, Robinson A, Rao K, Opfer E. Feasibility and acceptability of a diagnostic randomized clinical trial of bowel ultrasound in infants with suspected necrotizing enterocolitis. Eur J Pediatr. 2022 Aug;181(8):3211-3215. doi: 10.1007/s00431-022-04526-4. Epub 2022 Jun 17. PMID 35713688

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited based on gestational age and were only randomized into Arm A or Arm B upon suspicion of NEC. A total of 56 subjects were enrolled, but only 14 subjects were randomized to Arm A (n=8) or Arm B (n=6)
Period: Overall Study
Arm/Group | Arm A: AXR Only | Arm B: AXR + Bowel US
Started | 8 | 6
Completed | 8 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: AXR Only | Arm B: AXR + Bowel US | Total
Number analyzed (Participants) | 8 | 6 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8 | 6 | 14
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Standard Deviation); unit: Weeks] | 27.13 (2.03) | 26.50 (3.02) | 26.62 (2.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 1 | 7
  Male | 2 | 5 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 6 | 6 | 12
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 3 | 3
  White | 6 | 2 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 6 | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Requiring Medical Management
Description: Evaluate the difference between medical and surgical management between study arms.
  Medical management is defined as subjects whom did not undergo surgery for their NEC diagnosis.
  Surgical management is defined as subjects that had a surgical intervention for the NEC diagnosis.
  Please note that the study was terminated due to low enrollment numbers, thus statistically relevant and applicable numbers cannot be generated from this small study sample.
Time Frame: First 12 months
Measure: Number; unit: participants
Arm/Group | Arm A: AXR Only | Arm B: AXR + Bowel US
Number analyzed (Participants) | 8 | 6
participants | 1 | 1

2. Primary Outcome: Number of Days Between NEC Diagnosis and Surgical Intervention
Description: The number of days between NEC diagnosis and surgical intervention for those that need it. Days were continuously counted until subject was discharged from the hospital.
  Please note that the study was terminated due to low enrollment numbers, thus statistically relevant and applicable numbers cannot be generated from this small study sample.
Time Frame: 12 months
Population: Only two subjects underwent surgical intervention for their NEC diagnosis. One subject underwent surgery on the same day of diagnosis and the other subject 20 days after diagnosis.
Measure: Mean (95% Confidence Interval); unit: Days
Arm/Group | Arm A: AXR Only | Arm B: AXR + Bowel US
Number analyzed (Participants) | 0 | 2
Days |  | 10 [0 to 20]

3. Primary Outcome: Number of NPO Days
Description: Number of nothing by mouth (NPO) days between subject diagnosis of NEC to when subject was placed back on continuous feeds.
  Please note that the study was terminated due to low enrollment numbers, thus statistically relevant and applicable numbers cannot be generated from this small study sample.
Time Frame: 12 months
Population: Number of NPO days were evaluated from time of NEC diagnosis to when subject was placed back on continuous feeds.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Arm A: AXR Only | Arm B: AXR + Bowel US
Number analyzed (Participants) | 8 | 6
Days | 4 (3.6) | 7 (1.6)

ADVERSE EVENTS:
Time Frame: 22 months
Description: Participants were not at risk for an SAE, All-Cause Mortality or AE's due to the minimal risk nature of the study.
  Time Frame is expressed as the specific duration of time over which each participant was assessed from baseline forward.
Arm/Group | Arm A: AXR Only | Arm B: AXR + Bowel US
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8

LIMITATIONS AND CAVEATS:
Please note that the study was terminated due to low enrollment numbers, thus statistically relevant and applicable numbers cannot be generated from this small study sample.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-02-26): https://cdn.clinicaltrials.gov/large-docs/11/NCT03963011/Prot_SAP_002.pdf
  • Informed Consent Form (2020-05-20): https://cdn.clinicaltrials.gov/large-docs/11/NCT03963011/ICF_001.pdf